CLINICAL TRIAL: NCT01323439
Title: Axium™ MicroFX™ for Endovascular Repair of IntraCranial Aneurysm-A Multicenter Study
Acronym: AMERICA
Status: Completed | Type: Observational
Sponsor: Medtronic Neurovascular Clinical Affairs (Industry)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: AMERICA
Record Dates: First submitted 2011-03-23; First posted 2011-03-25 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Aneurysm
Keywords: Patients presenting with an intracranial aneurysm
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Axium™ MicroFX™ PGLA Treated Subjects: This observational evaluation will evaluate early experience using the Axium™ MicroFX™ PGLA COILS as compared to published literature of coils with electrolytic, thermal or hydraulic detachment process or the Axium™ Bare Detachable Coils arm obtained from previous evaluation conducted following the same protocol
  Interventions: Device: Axium™ MicroFX™ PGLA COILS

INTERVENTIONS:
Device: Axium™ MicroFX™ PGLA COILS — Axium™ MicroFX™ PGLA COILS to treat aneurysms

SUMMARY:
This is a multicenter, prospective single-arm trial evaluating the safety and efficacy of the Axium MicroFX coil system in 100 aneurysms.

DETAILED DESCRIPTION:
This is a multicenter, prospective single-arm trial evaluating the safety and efficacy of the Axium MicroFX coil system in 99 patients at 13 study centers. The primary endpoint of the trial was the anatomic occlusion of the aneurysm in the immediate post-procedure angiogram basedon the Raymond classification. Secondary endpoints included safety during the procedure, safety after the procedure, detachment system performance, stability of the embolization, and packing efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of one or more intracranial aneurysm, either ruptured or unruptured.
* Information on data collection provided to the patient or legally authorized representative and signed informed consent.
* Aneurysm diameter ≤10mm .
* Age range of 18 - 90.

Exclusion Criteria:

* Aneurysm previously treated.
* Aneurysm AVM related or dissecting.
* Participation in a clinical investigation of other aneurysm treating or related devices.
* Any condition that would preclude the conduct of protocol follow-up.
* Aneurysm anatomy that is determined inappropriate for Axium coil placement, prior to opening of an Axium coil.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting with an intracranial aneurysm will be evaluated by the neuro interventional team, in accordance with institutional practice, to establish an appropriate treatment plan based on the patient's medical condition and available diagnostic screening prior to recruitment
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2010-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Anatomic occlusion of the aneurysm | Immediately post-procedure
  Occlusion of aneurysm based on the Raymond classification

SECONDARY OUTCOMES:
Safety during the procedure | Discharge, up to two years
  Morbidity and mortality rate
Safety post-procedure | 3-6 months follow-up
  Morbidity and mortality rate
Detachment system performance | During procedure
  Occurrence of detachment failure
Stability of embolization | 3-6 months follow-up
  Rate of change towards worsening Raymond grades
Packing efficacy | 36- months follow-up
  increase in packing density calculated as ration between volume of coils and the aneurysm volume

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No